CLINICAL TRIAL: NCT00562796
Title: Prevalence and Metabolic Consequences of Relative Growth Hormone Deficiency in Abdominal Obesity
Brief Title: Prevalence and Cardiovascular Effects of Growth Hormone Deficiency in Abdominal Obesity
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 555; 1R01HL085268-01A1 (NIH)
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Obesity; Growth Hormone
Keywords: Growth Hormone Deficiency; Cardiovascular Disease; Intra-abdominal Fat; Insulin Resistance
MeSH Terms: conditions — Obesity; Dwarfism, Pituitary; Cardiovascular Diseases; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples will include serum, plasma, whole blood, and white blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Participants with abdominal obesity without growth hormone deficiency
- 2: Participants with abdominal obesity with growth hormone deficiency
- 3: Participants who are lean controls

SUMMARY:
Obesity is one of the leading causes of cardiovascular-related diseases, including diabetes and heart disease. Obesity, and more specifically abdominal obesity, may cause decreased growth hormone (GH) levels. It is believed that GH deficiency may contribute to increased cardiovascular risk by affecting insulin resistance, inflammatory markers, and blood cholesterol levels. This study will determine the occurrence of GH deficiency in abdominal obesity and whether GH deficiency is associated with increased cardiovascular risk beyond traditional risk factors.

DETAILED DESCRIPTION:
Obesity is associated with significant morbidity and mortality and is a primary public health concern. Both the incidence and prevalence of obesity have increased over the last several decades, with obesity now affecting an estimated 31% of the American population. Recent data suggest that people with abdominal obesity commonly exhibit low levels of GH, which affects the body's growth rate and the way the body uses food for energy. Low GH levels and excess abdominal fat have been linked to improper functioning of the cardiovascular system and, therefore, may increase one's risk of cardiovascular disease. This study will determine the prevalence of GH deficiency in abdominal obesity and whether GH deficiency is associated with increased cardiovascular risk beyond traditional risk factors.

Participation in this observational study will last between 2 and 4 weeks. The study will consist of two outpatient visits, held at either the Massachusetts General Hospital or Massachusetts Institute of Technology. Visit 1 will last 4 hours and will include a physical exam, medical history, blood draw, urine sampling, indirect calorimetry test, and growth hormone releasing hormone (GHRH)+Arginine stimulation test. Eligible participants will return within the next 3 weeks for Visit 2, which will last 5 hours. Before the second visit, participants will be asked to record their food intake for 4 days on a food record. During the visit, participants will have a repeat physical exam, urine sampling, and blood draw. Participants will also undergo an oral glucose tolerance test, whole body DEXA scan, abdominal computed tomography (CT) scan, and a carotid ultrasound. Participation in the study will end after Visit 2.

ELIGIBILITY:
Inclusion Criteria for Obesity:

* Body mass index (BMI) greater than or equal to 30 kg/m2
* Abdominal obesity, defined as waist circumference greater than or equal to 102 cm in men and greater than or equal to 88 cm in women

Inclusion Criteria for Lean Controls:

* BMI less than 25 kg/m2
* Waist circumference less than 102 cm in men and less than 88 cm in women

Exclusion Criteria for both groups:

* Obesity due to known secondary causes
* Taking any weight lowering drugs
* Previous bariatric surgery
* Use of the following compounds within the 3 months prior to study entry: estrogen, progesterone, GH, GHRH, glucocorticoids, megesterol acetate, antidiabetic agents, oral contraceptive pills, or any other hormone or drug known to affect GH levels
* Change in lipid lowering or antihypertensive regimen within 3 months prior to study entry
* Use of testosterone or hormone replacement therapy
* Previously known diabetes mellitus or other severe chronic illness
* Hemoglobin less than 11.0 g/dL, creatinine greater than 1.5 mg/dL, or serum glutamic oxaloacetic transaminase (SGOT) greater than 2.5 times the upper limit of normal
* Follicle stimulating hormone (FSH) greater than 20 IU/L in women
* Positive urine pregnancy test
* Prior history of pituitary disease, pituitary surgery, head irradiation, or any other condition known to affect the GH axis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will include participants from the community at large who are able to come to either the Massachusetts General Hospital (MGH) Weight Center or Massachusetts Institute of Technology for study visits.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of growth hormone deficiency | Measured at baseline

SECONDARY OUTCOMES:
Carotid intima-media thickness, visceral adiposity, glucose intolerance, inflammatory markers, mitochondrial function, physical activity and adipocytokines | Measured at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Grinspoon, MD, Principal Investigator — Program in Nutritional Metabolism, Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Stanley TL, Feldpausch MN, Murphy CA, Grinspoon SK, Makimura H. Discordance of IGF-1 and GH stimulation testing for altered GH secretion in obesity. Growth Horm IGF Res. 2014 Feb;24(1):10-5. doi: 10.1016/j.ghir.2013.11.001. Epub 2013 Nov 15. PMID 24291224
- [Derived] Makimura H, Feldpausch MN, Stanley TL, Sun N, Grinspoon SK. Reduced growth hormone secretion in obesity is associated with smaller LDL and HDL particle size. Clin Endocrinol (Oxf). 2012 Feb;76(2):220-7. doi: 10.1111/j.1365-2265.2011.04195.x. PMID 21819438
- [Derived] Makimura H, Stanley TL, Sun N, Connelly JM, Hemphill LC, Hrovat MI, Systrom DM, Grinspoon SK. Increased skeletal muscle phosphocreatine recovery after sub-maximal exercise is associated with increased carotid intima-media thickness. Atherosclerosis. 2011 Mar;215(1):214-7. doi: 10.1016/j.atherosclerosis.2010.11.037. Epub 2010 Dec 5. PMID 21185022
- [Derived] Makimura H, Stanley TL, Sun N, Connelly JM, Hemphill LC, Grinspoon SK. The relationship between reduced testosterone, stimulated growth hormone secretion and increased carotid intima-media thickness in obese men. Clin Endocrinol (Oxf). 2010 Nov;73(5):622-9. doi: 10.1111/j.1365-2265.2010.03859.x. PMID 20681993
- [Derived] Makimura H, Stanley T, Mun D, Chen C, Wei J, Connelly JM, Hemphill LC, Grinspoon SK. Reduced growth hormone secretion is associated with increased carotid intima-media thickness in obesity. J Clin Endocrinol Metab. 2009 Dec;94(12):5131-8. doi: 10.1210/jc.2009-1295. Epub 2009 Oct 16. PMID 19837914